CLINICAL TRIAL: NCT05215795
Title: Validity and Reliability of Modified Box and Block Test and Targeted Box and Block Test in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Lecturer, MSc PT, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU3
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Validity; Reliability; Modified Box and Block Test; Targeted Box and Block Test; Upper Extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is investigated validity and reliabilty of Modified Box and Block Test and Targeted Box and Block Test in patients with stroke.

DETAILED DESCRIPTION:
Fifty patients with stroke will included in the study. Box and Block Test, Modified Box and Block Test, Targeted Box and Block Test, 9 Hole Peg Test, Fugl-Meyer Assessment of the upper extremity will used to assess upper extremity. To evaluate validity between Modified and Targeted Box and Block Tests and Box and Block Test, 9 Hole Peg Test, Fugl-Meyer Assessment will used to correlation analysis tests. The investigator will evaluate after one week to test-retest reliability to patients. Other pyhsiotherapist will evaluate to patients inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke and in the chronic phase (having been diagnosed with stroke at least 6 months ago),
* Over 18 years old,
* Mini Mental Test score ≥ 24 points,
* Able to grasp and release a 2.5 cm cube on both upper extremities,
* Brunnstrom Upper Extremity Staging ≥ 3
* Modified Ashworth Scale ≤ 2,
* Able to sit independently in a chair for 2 minutes

Exclusion Criteria:

* Having a neurological disease other than stroke
* Have had surgery in the last 6 months
* Severely affected upper extremity
* Uncooperative with physiotherapist
* Patients with neglect, aphasia and hemianopsia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Modified Box and Block Test | 10 minute
  The Modified Box and Block (mBBT) test is an upper extremity performance test.Unlike BBT, in mBBT, instead of randomly picking the cubes, 16 cubes are arranged in a certain order.
  The cubes are asked to take the other cubes in that row, starting from the innermost left cube, first to the right, and then to the next upper row.
  It is recorded how many seconds passed through 16 cubes placed at a certain level.
Targeted Box and Block Test | 10 minute
  In tBBT, as in mBBT, the time of passing 16 cubes over the obstacle to the other side is recorded. However, the difference from mKBT is that 16 cubes are placed at a certain level, but the patients are asked to place the cubes on the other side in 4 cm squares where the cube will be placed.
  These squares correspond to the left symmetrical position of the cube on the right.
  In this way, patients have to place the cube they grasp only at the desired point.

SECONDARY OUTCOMES:
9 Hole Peg Test | 10 minute
  9HPT is a dexterity test.The patient is asked to place the 9 wooden blocks into the 9 holes in the maximum amount of time.Then he is asked to take it out and put it back in its place. The total time is recorded.
Fugl-Meyer Assessment for Upper Extremity | 15 minutes
  The Fugl-Meyer Assessment is a disease-specific impairment index designed to assess motor function, balance, sensation qualities and joint function in hemiplegic post-stroke patients.The scale consists of four categories (Shoulder/Elbow/Forearm, Wrist, Hand/Finger, and Coordination) and evaluates 23 different movements in 33 sections.The maximum score is 66 points
Box and Block Test | 5 minute
  Box and Block (mBBT) test is an upper extremity performance test. The patient is instructed to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds. The number of cubes passed to the other side in 60 seconds is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye AKKURT, MSc, Principal Investigator — Kutahya Health Sciences University; Cihan Caner AKSOY, PhD, Study Director — Kutahya Health Sciences University; Fatıma YAMAN, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)